CLINICAL TRIAL: NCT02766036
Title: Propolis Effects on Proteinuria and Kidney Function in Patients With Chronic Kidney Disease
Brief Title: Propolis Effects in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcelo Augusto Duarte Silveira, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54326916.4.0000.0068; USP Brazil (Other: University of São Paulo School of Medicine)
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Proteinuria; Propolis; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis (Active Comparator): Patients will continue to receive standard treatment for their comorbidities, determined by the attending physician. Patients will receive 500 mg / day of the propolis extract in the form of tablets split in two daily doses.
  Interventions: Drug: Propolis
- Placebo (Placebo Comparator): Patients will continue to receive standard treatment for their comorbidities, determined by the attending physician. Patients will receive 500 mg / day of the propolis-placebo in the form of tablets split in two daily doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propolis — Patients will receive 500 mg / day of the propolis extract in the form of tablets split in two daily doses
  Arms: Propolis
Drug: Placebo — Patients will receive 500 mg / day of the placebo in the form of tablets split in two daily doses
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the impact of Propolis on proteinuria reduction and protection of the glomerular filtration rate in chronic renal failure patients.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years;
* less than 90 years;
* glomerular filtration rate between 25 and 70 ml / min;
* proteinuria in the urine 24 hours more than 300 mg or protein / creatinina in isolated urine greater than 0.3g / g or microalbuminuria (albumin / creatinine ratio) between 30-300 mg / g.

Exclusion Criteria:

* Pregnants;
* Neoplasia carrier;
* Renal transplant patients;
* Patients who refuse to participate in the study.
* Glomerulopathy on Immunosuppression

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Reducing Proteinuria | One year
  Reduction from baseline proteinuria.

SECONDARY OUTCOMES:
Protection of the glomerular filtration rate | One year
  Maintaining glomerular filtration rate or inferior reduction to 5 ml per minute per 1.73 m2 of body-surface area from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: General Hospital, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be evaluated monthly by researchers at the scientific meetings of the department. Data from this study will be considered joint property of the parties involved. Researchers are, however, responsible for committing to make public the results.
Supporting Information: Study Protocol
Time Frame: The results of this research will be published to become public domain.

REFERENCES:
- [Background] Fujihara CK, DE Lourdes Noronha I, Malheiros DMAC, Antunes GR, DE Oliveira IB, Zatz R. Combined mycophenolate mofetil and losartan therapy arrests established injury in the remnant kidney. J Am Soc Nephrol. 2000 Feb;11(2):283-290. doi: 10.1681/ASN.V112283. PMID 10665935
- [Background] da Costa MF, Liborio AB, Teles F, Martins Cda S, Soares PM, Meneses GC, Rodrigues FA, Leal LK, Miron D, Silva AH, Martins AM. Red propolis ameliorates ischemic-reperfusion acute kidney injury. Phytomedicine. 2015 Aug 15;22(9):787-95. doi: 10.1016/j.phymed.2015.03.017. Epub 2015 Apr 12. PMID 26220625
- [Result] Teles F, da Silva TM, da Cruz Junior FP, Honorato VH, de Oliveira Costa H, Barbosa AP, de Oliveira SG, Porfirio Z, Liborio AB, Borges RL, Fanelli C. Brazilian red propolis attenuates hypertension and renal damage in 5/6 renal ablation model. PLoS One. 2015 Jan 21;10(1):e0116535. doi: 10.1371/journal.pone.0116535. eCollection 2015. PMID 25607548
- [Result] Machado JL, Assuncao AK, da Silva MC, Dos Reis AS, Costa GC, Arruda Dde S, Rocha BA, Vaz MM, Paes AM, Guerra RN, Berretta AA, do Nascimento FR. Brazilian green propolis: anti-inflammatory property by an immunomodulatory activity. Evid Based Complement Alternat Med. 2012;2012:157652. doi: 10.1155/2012/157652. Epub 2012 Dec 19. PMID 23320022
- [Result] Himmelfarb J. Linking oxidative stress and inflammation in kidney disease: which is the chicken and which is the egg? Semin Dial. 2004 Nov-Dec;17(6):449-54. doi: 10.1111/j.0894-0959.2004.17605.x. PMID 15660575
- [Result] Inker LA, Coresh J, Levey AS, Tonelli M, Muntner P. Estimated GFR, albuminuria, and complications of chronic kidney disease. J Am Soc Nephrol. 2011 Dec;22(12):2322-31. doi: 10.1681/ASN.2010111181. Epub 2011 Sep 30. PMID 21965377
- [Result] Shah SV, Baliga R, Rajapurkar M, Fonseca VA. Oxidants in chronic kidney disease. J Am Soc Nephrol. 2007 Jan;18(1):16-28. doi: 10.1681/ASN.2006050500. Epub 2006 Dec 13. PMID 17167116
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Silveira MAD, Teles F, Berretta AA, Sanches TR, Rodrigues CE, Seguro AC, Andrade L. Effects of Brazilian green propolis on proteinuria and renal function in patients with chronic kidney disease: a randomized, double-blind, placebo-controlled trial. BMC Nephrol. 2019 Apr 25;20(1):140. doi: 10.1186/s12882-019-1337-7. PMID 31023272